CLINICAL TRIAL: NCT04946305
Title: A Post Marketing Surveillance on Lutathera® (Lutetium (177Lu) Oxodotreotide, 177Lu-DOTA0-Tyr3-Octreotate) in Patients With Somatostatin Receptor Positive Gastroenteropancreatic Neuroendocrine Tumor (GEP-NET) in Korea
Brief Title: A Post Marketing Surveillance on Lutathera® in Patients With Somatostatin Receptor Positive Gastroenteropancreatic Neuroendocrine Tumor in Korea
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAAA601A12403
Record Dates: First submitted 2021-06-23; First posted 2021-06-30 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Somatostatin Receptor-positive GEP-NET
Keywords: somatostatin receptor-positive GEP-NET; Lutathera; Observational; prospective
MeSH Terms: interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lutathera: Patients administered Lutathera by prescription
  Interventions: Other: Lutathera

INTERVENTIONS:
Other: Lutathera — Prospective observational study. There is no treatment allocation. Patients administered Lutathera by prescription that have started before inclusion of the patient into the study will be enrolled.

SUMMARY:
This is a prospective, open-label, multi-center, non-comparative, non-interventional observational study to assess safety and effectiveness of Lutathera in patients with somatostatin receptor-positive GEP-NET in the real-world setting in Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who start Lutathera treatment per clinical judgment, according to the locally approved labeling.

   - somatostatin receptor-positive gastroenteropancreatic neuroendocrine tumors (GEP-NETs) in adults.
2. Patients who are willing to provide written informed consent.

Exclusion Criteria:

1. Patients with contraindication according to prescribing information for Lutathera in Korea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with somatostatin receptor-positive GEP-NET in the real-world setting in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 36 weeks
  Incidence of Adverse Events (AEs), Serious AE and unexpected AEs.
Incidence of Adverse Drug Reactions | Up to 36 weeks
  Incidence of Adverse Drug Reactions (ADRs), Serious ADRs and unexpected ADRs.

SECONDARY OUTCOMES:
Effectiveness in terms of Overall Response Rate (ORR) | Up to 32 weeks (4 cycles of 8 weeks)
  ORR is defined as the proportion of treated patients who achieve a best overall response of partial response (PR) or complete response (CR) according to RECIST 1.1.
  Partial Response (PR): At least a 30% decrease from baseline, confirmed at 4 weeks.
  Complete Response (CR): Disappearance of all known disease, confirmed at 4 weeks, lymph nodes must be less than 10 mm short axis

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- South Korea (2):
  - Novartis Investigative Site, Seongnam-si, Gyeonggi-do
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No